CLINICAL TRIAL: NCT06493656
Title: The Efficacy of Single-shot Capsule-preserving Hydrodilatation With Corticosteroids in Treating Adhesive Capsulitis of the Shoulder: A Randomized Controlled Trial Versus Isolated Corticosteroid Injection
Brief Title: Isolated Glenohumeral Corticosteroid Injection Versus Concomitant Capsule Preserving Hydrodilatation
Acronym: CSvsCSHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Jung-Taek Hwang, Professor, Chuncheon Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSvsCSHD
Record Dates: First submitted 2024-06-24; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Adhesive Capsulitis; Adhesive Capsulitis of Shoulder
Keywords: Glenohumeral injection; Hydrodilatation; Corticosteroid injection
MeSH Terms: conditions — Bursitis | interventions — Adrenal Cortex Hormones; Triamcinolone; Lidocaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Study group underwent ultrasound-guided posterior approach of glenohumeral space injection for adhesive capsulitis of the shoulder. The injection mixture was: 1 mL triamcinolone, 4 mL lidocaine, 7 mL normal saline.
  Control group underwent ultrasound-guided posterior approach of glenohumeral space HYDRODILATATION for adhesive capsulitis of the shoulder. The injection mixture was: 1 mL triamcinolone, 4 mL lidocaine, 15 mL normal saline.
Who Masked: Participant, Outcomes Assessor
Masking Description: A final number of 50 patients were enrolled in the trial and randomly assigned to either the isolated corticosteroid injection group (Group CS) or the concomitant hydrodilatation group (Group CSHD). Double-blinded randomization was performed by an independent nurse using a computer-generated random sequence. A musculoskeletal radiologist, blinded to group allocation, performed the diagnostic ultrasound and MRI interpretations. A blinded orthopaedic nurse carried out the physical examination and clinical scoring.
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- Isolated corticosteroid injection (Experimental): Ultrasound-guided posterior approach of glenohumeral space injection for adhesive capsulitis of the shoulder. The injection mixture was: 1 mL triamcinolone, 4 mL lidocaine.
  Interventions: Procedure: Ultrasound-guided glenohumeral space isolated corticosteroid injection; Drug: 1mL of Triamcinolone (40mg/1mL) Injectable Solution; Drug: 4mL of Lidocaine 1% Solution Injectable Solution
- Concomitant hydrodilatation with corticosteroid injection (Active Comparator): Ultrasound-guided posterior approach of glenohumeral space hydrodilatation for adhesive capsulitis of the shoulder. The injection mixture was: 1 mL triamcinolone, 4 mL lidocaine, and 15 mL normal saline
  Interventions: Procedure: Ultrasound-guided glenohumeral space concomitant hydrodilatation with corticosteroid injection; Drug: 1mL of Triamcinolone (40mg/1mL) Injectable Solution; Drug: 4mL of Lidocaine 1% Solution Injectable Solution; Drug: 15mL of Normal Saline

INTERVENTIONS:
Procedure: Ultrasound-guided glenohumeral space isolated corticosteroid injection — Using a 21-gauge spinal needle, the predefined steroid solution was injected under ultrasound guidance using 5- to 13-MHz linear probe into the glenohumeral space through the posterior approach.
  Arms: Isolated corticosteroid injection
Procedure: Ultrasound-guided glenohumeral space concomitant hydrodilatation with corticosteroid injection — Using a 21-gauge spinal needle, the predefined steroid solution with additional 15 mL of normal saline was injected under ultrasound guidance using 5- to 13-MHz linear probe into the glenohumeral space through the posterior approach.
  Arms: Concomitant hydrodilatation with corticosteroid injection
Drug: 1mL of Triamcinolone (40mg/1mL) Injectable Solution — 1mL of Triamcinolone 40mg/1mL solution was included in the injection/hydrodilatation regimen.
Drug: 4mL of Lidocaine 1% Solution Injectable Solution — 4mL of 1% Lidocaine solution was included in the injection/hydrodilatation regimen.
Drug: 15mL of Normal Saline — 15mL of 1% Lidocaine solution was included in the hydrodilatation regimen.
  Arms: Concomitant hydrodilatation with corticosteroid injection

SUMMARY:
This clinical trial investigates whether concomitant capsule-preserving hydrodilatation (CSHD) is more effective than isolated glenohumeral corticosteroid injection (CS) in treating shoulder adhesive capsulitis. The main questions it aims to answer are

* Is CSHD inferior to CS in immediate pain relief as the solution is diluted?
* Is CSHD superior to CS in improving the range of motion as the contracted capsule is dilated?

Group CS will receive an ultrasound-guided glenohumeral corticosteroid injection only, with a solution of 5 mL.

Group CSHD will receive an ultrasound-guided glenohumeral corticosteroid with hydrodilatation, with a solution of 20 mL.

Clinical scores and range of motion will be compared between the groups up to six months post-injection.

DETAILED DESCRIPTION:
A single-centre, double-blinded, prospective randomised controlled trial involving patients diagnosed with adhesive capsulitis of the shoulder (AC).

Patients were randomly allocated to either corticosteroid injection with hydrodilatation (group CSHD) or corticosteroid injection only (group CS).

For the CS group, a solution of 1 mL triamcinolone (40mg) and 4 mL 1% lidocaine, 5 mL in total, was injected intraarticularly through the posterior approach using ultrasound guidance.

The CSHD group received an injection of 20 mL with 15 mL of normal saline added to the abovementioned 5 mL solution. The dilatation of the joint capsule was confirmed by the increase in distance between the capsule and the humeral head.

Patients underwent the following assessments just before the injection, and at post-injection three weeks, seven weeks, three months, and six months.

Range of motion in forward elevation, external rotation, and internal rotation Clinical scores include the pain visual analogue scale (pVAS), the American Shoulder and Elbow Surgeons score, and the Constant-Murley score.

Subjective patient satisfaction was recorded on a scale from 0 to 100, with 100 being the most satisfied.

The recorded data were compared within each group before and after the injection, and also between the groups.

ELIGIBILITY:
Inclusion Criteria:

Two or more of the following criteria within the shoulder's range of motion:

* Abduction and forward elevation below 100˚
* External rotation at the side below 30˚
* Internal rotation at 90˚ of abduction below 30˚

Exclusion Criteria:

* History of shoulder surgery, trauma, nerve injury
* Concomitant rotator cuff/biceps lesions in ultrasound or MRI
* Glenohumeral arthritis in simple X-ray
* Calcific tendinosis in simple X-ray
* Underlying conditions: cancer, mental illness, hormonal imbalance
* Diabetes with HbA1c levels exceeding 7.0%

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-12-05 (Actual); Primary Completion 2015-11-17 (Actual); Study Completion 2015-11-17 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) for pain | Change from the baseline to 6 months
  Patient-reported 0-10 scale of pain, 0: no pain, 10: very severe pain

SECONDARY OUTCOMES:
Range of motion (ROM) | Change from the baseline to 6 months
  ROM in degrees, forward elevation (0-150), external rotation (0-90), and internal rotation (0-90)
American Shoulder and Elbow Surgeons (ASES) shoulder score | Change from the baseline to 6 months
  Patient-reported shoulder satisfaction score, 0-100, higher scores mean a better outcome.
Constant-Murley score | Change from the baseline to 6 months
  Patient-reported and healthcare provider-assessed shoulder satisfaction score, 0-100, higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jung Taek Hwang, MD, PhD, Principal Investigator — Chuncheon Sacred Heart Hospital
Locations (1):
- Chuncheon Sacred Heart Hospital, Chuncheon, Gangwondo, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Neviaser AS, Hannafin JA. Adhesive capsulitis: a review of current treatment. Am J Sports Med. 2010 Nov;38(11):2346-56. doi: 10.1177/0363546509348048. Epub 2010 Jan 28. PMID 20110457
- [Result] Cho CH, Lee YH, Kim DH, Lim YJ, Baek CS, Kim DH. Definition, Diagnosis, Treatment, and Prognosis of Frozen Shoulder: A Consensus Survey of Shoulder Specialists. Clin Orthop Surg. 2020 Mar;12(1):60-67. doi: 10.4055/cios.2020.12.1.60. Epub 2020 Feb 13. PMID 32117540
- [Result] Redler LH, Dennis ER. Treatment of Adhesive Capsulitis of the Shoulder. J Am Acad Orthop Surg. 2019 Jun 15;27(12):e544-e554. doi: 10.5435/JAAOS-D-17-00606. PMID 30632986
- [Result] Catapano M, Mittal N, Adamich J, Kumbhare D, Sangha H. Hydrodilatation With Corticosteroid for the Treatment of Adhesive Capsulitis: A Systematic Review. PM R. 2018 Jun;10(6):623-635. doi: 10.1016/j.pmrj.2017.10.013. Epub 2017 Nov 10. PMID 29129609
- [Result] Oh JH, Oh CH, Choi JA, Kim SH, Kim JH, Yoon JP. Comparison of glenohumeral and subacromial steroid injection in primary frozen shoulder: a prospective, randomized short-term comparison study. J Shoulder Elbow Surg. 2011 Oct;20(7):1034-40. doi: 10.1016/j.jse.2011.04.029. Epub 2011 Aug 4. PMID 21816628
- [Result] Kim DY, Lee SS, Nomkhondorj O, Cho MG, Lee JJ, Hwang JT, Hong MS. Comparison Between Anterior and Posterior Approaches for Ultrasound-Guided Glenohumeral Steroid Injection in Primary Adhesive Capsulitis: A Randomized Controlled Trial. J Clin Rheumatol. 2017 Jan;23(1):51-57. doi: 10.1097/RHU.0000000000000475. No abstract available. PMID 28002160